CLINICAL TRIAL: NCT01034787
Title: Open Label Phase II Study of AntiCTLA4 in Patients With Unresectable or Metastatic Uveal Melanoma
Brief Title: Study of AntiCTLA4 in Patients With Unresectable or Metastatic Uveal Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Principal Investigator, Tina Cheng, Dr. Tina Cheng, AHS Cancer Control Alberta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBCC 905001
Record Dates: First submitted 2009-12-15; First posted 2009-12-17 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Uveal Melanoma
Keywords: CP-675,206; Immunotherapy; AntiCTLA4; Clinical Trial; Unresectable or Metastatic
MeSH Terms: conditions — Uveal Melanoma; Neoplasm Metastasis | interventions — tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open Label CP-675,206 (Experimental): Patients will receive CP-675,206 at 15 mg/kg administered intravenously on day 1 of every 90-day cycle for up to 4 cycles or until disease progression or intolerance of toxicity.
  Interventions: Drug: CP-675,206

INTERVENTIONS:
Drug: CP-675,206 — Patients will receive CP-675,206 at 15 mg/kg administered intravenously on day 1 of ever 90 cycle for up to 4 cycles or until progression or intolerance of toxicity. Tumor assessments will be done ever 3 months. Additional scans will be done if clinically indicated.

SUMMARY:
This is a Phase 2, multi-center, open-label study in patients with surgically incurable stage III or IV uveal melanoma who have not received prior immunotherapy. CP-675,206 is thought to stimulate patients' immune systems to attack their tumors. CP-675,206 has been shown to induce durable tumor responses in patients with metastatic melanoma in phase 1 and phase 2 clinical studies.

DETAILED DESCRIPTION:
This is a Phase 2, multi-center, open-label study in patients with surgically incurable stage III or IV uveal melanoma who have not received prior immunotherapy. Patients may have received prior chemotherapy or biological therapy for the treatment of advanced disease. Twenty-nine patients will be enrolled. Patients may have either measurable disease or non-measurable disease.

Patients will receive CP-675,206 at 15 mg/kg administered intravenously on day 1 of every 90-day cycle for up to 4 cycles or until disease progression or intolerance of toxicity. Each cycle is defined as a 90 +/- 4 days period. Patients should be weighed within 10 days prior to each cycle and the administered dose of CP-675,206 should be recalculated.

Patients who complete 4 doses of CP-675,206 without disease progression and who subsequently experience disease progression more than 3 months after the last dose may receive 4 additional doses of CP-675,206 provided that they have not received other systemic therapy for their melanoma. Patients with clinical benefit may be considered for additional dosing if evidence emerges supporting ongoing maintenance therapy.

Tumor assessments will be done every 3 months. All patients with objective tumor response must have additional scans scheduled 4-6 weeks after the criteria for response are first met in order to confirm the response. Additional scans will be done if clinically indicated. Survival will be monitored on all patients for up to 5 years from the date of first dose of CP-675,206. The follow up time may be adjusted based on ongoing studies using CP-675,206 for melanoma.

An exploratory study will be conducted to identify micro environmental features in the tumor that are permissive of tumor immunity (i.e: those associated with a "response" to anti-CTLA4) and to assess whether anti-CTLA4 causes peripheral mobilization of immunomodulatory inflammatory cells.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed uveal melanoma including choroidal melanoma, iris melanoma, and ciliary body melanoma
* Patients may either have measurable disease or non-measurable disease.
* Biopsies from a readily accessible site of disease on study enrollment are mandatory in principle. Waivers will be granted if there are no accessible lesions. The collection of a representative block of the diagnostic tumour tissue (if available) is mandatory.
* ECOG performance status of 0 or 1
* Age 18 years or older
* Adequate bone marrow, hepatic, and renal function determined within 14 days prior to registration, defined as:
* Serum lactic acid dehydrogenase (LDH) </= 1.5 x ULN.
* Alkaline phosphatase (ALP) </= 2 x ULN.
* No weight loss >/= 10% in the proceeding 4 weeks.
* CT scan of the brain with contrast or MRI of the brain within 28 days of registration showing no evidence of brain metastases.
* Females of childbearing potential must have a negative serum or urine pregnancy test within 14 days prior to registration. Females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential.
* Females of childbearing potential and males who have not undergone surgical sterilization must agree to practice a form of effective contraception prior to entry into the study and for 12 months following the last dose of study drug. The definition of effective contraception will be based on the judgment of the investigator.

Exclusion Criteria:

* Melanoma of cutaneous, mucosal or conjunctival origin.
* History of brain or leptomeningeal metastases.
* Received any prior CTLA4 inhibiting agent (eg MDX-010, ipilimumab) or other immunotherapy.
* History of chronic inflammatory or autoimmune disease
* History of uveitis or melanoma-associated retinopathy.
* History of inflammatory bowel disease, celiac disease, or other chronic gastrointestinal conditions associated with diarrhea or bleeding, or current acute colitis of any origin.
* History of hepatitis due to Hepatitis B virus or Hepatitis C virus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-08-17 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2017-08-08 (Actual)

PRIMARY OUTCOMES:
Progression-free survival at 6 months after initiation of CP-675,206 | 6 months
  A 6-month progression free survivor will be defined as a patient who is alive and who has not progressed at 6 months or more post treatment.

SECONDARY OUTCOMES:
Objective tumor response | overall
  Duration of Objective response (CR or PR) for responding patients will be measured from the date of registration to the date of progression or death due to progressive disease, whichever occurs first. In addition, the Duration of Complete Response will be measured from the date that a CR was first documented to the date of progression or death due to progressive disease, whichever occurs first.
Durable response | 6 or more months
  Durable response is defined as an objective tumor response that last 6 or more months
Median survival and overall survival | overall
  • Overall Survival (OS) is defined as the time from the date of registration to date of death by any cause. In the absence of confirmation of death, survival time will be censored at the last date the patient was known to be alive.
Adverse events and tolerability | overall
  Following the first dose, adverse events should be continuously assessed and documented during the study reporting period. Adverse events will be followed up to and including the End of Treatment visit. Additionally, all adverse events with a causal relationship to the study drug must be followed until the event and its sequalae have resolved, returned to baseline, been deemed irreversible, or until the patient dies.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Background] Rietschel P, Panageas KS, Hanlon C, Patel A, Abramson DH, Chapman PB. Variates of survival in metastatic uveal melanoma. J Clin Oncol. 2005 Nov 1;23(31):8076-80. doi: 10.1200/JCO.2005.02.6534. PMID 16258106
- [Background] Bedikian AY, Legha SS, Mavligit G, Carrasco CH, Khorana S, Plager C, Papadopoulos N, Benjamin RS. Treatment of uveal melanoma metastatic to the liver: a review of the M. D. Anderson Cancer Center experience and prognostic factors. Cancer. 1995 Nov 1;76(9):1665-70. doi: 10.1002/1097-0142(19951101)76:93.0.co;2-j. PMID 8635073